CLINICAL TRIAL: NCT00287027
Title: Family Perspectives:Treatment of Psychiatric Illnesses With Atypical Long Acting Injectable Antipsychotic Medication
Status: Terminated | Type: Observational
Sponsor: National Alliance on Mental Illness New Hampshire (Other)
Collaborators: Janssen Medical Affairs (Industry)
Other Study IDs: CPHS#17558
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Psychotic Disorders
Keywords: psychotic disorders; family burden; long acting injectible antipsychotic medication
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Risperdal Long Acting Injectable Antipsychotic Medication

SUMMARY:
Patients who have schizophrenia, schizoaffective disorder, a psychotic disorder, and are being treated with a medication called Risperidone Long Acting Injectable medication or another antipsychotic medication are candidates for the study. The purpose of the study is to find out from patients' family how they feel the medication has affected their relationship with them. The study will involve meeting with family members three times over the course of one year. The first time will be at New Hampshire Hospital (NHH) or at a community mental health center and the follow up times will be at a convenient place and time for the family member (s), in the community. We will ask them to answer questions from the Family Burden Interview and Quality of Life Questionnaire. The family will not be charged for any test that is completed solely for this study. The family will be provided a travel stipend to meet with the researchers.

DETAILED DESCRIPTION:
Patients who have schizophrenia, schizoaffective disorder, a psychotic disorder, and are being treated with a medication called Risperidone Long Acting Injectable medication or another antipsychotic medication are candidates for the study. The purpose of the study is to find out from patients' family how they feel the medication has affected their relationship with them.The study will involve meeting with family members three times over the course of one year. The first time will be at New Hampshire Hospital (NHH) or at a community mental health center and the follow up times will be at a convenient place and time for the family member (s), in the community. We will ask them to answer questions from the Family Burden Interview and Quality of Life Questionnaire. The family will not be charged for any test that is completed solely for this study. The family will be provided a travel stipend to meet with the researchers.We do not see that there will be any risks to the family. We will be interviewing the patient's family, and they will be sharing information as to how they feel their relationship with the patient is going. All efforts will be made to keep this information confidential; however, there may be unforeseen circumstances that could lead to breaching of confidentiality. If the family expresses need for help the research staff will make recommendations for referral to a provider.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:Families of adults between the ages of 18-65 who have a diagnosis of Schizophrenia, Schizoaffective Disorder, Psychotic Disorder NOS, and whose loved one gave permission for them to be contacted.

* Either a) a family member whose adult consumer started on Risperidone Long Acting Injection within one month, while at New Hampshire Hospital and/or at a Community Mental Health Center and who consented to participate; or b) a family member whose adult consumer was switched from one antipsychotic medication to another (excluding clozapine) within one month, while at New Hampshire Hospital and/or at a Community Mental Health Center and who consented to participate.
* Families that have at least 4 hours per week contact with their loved one with mental illness for 2 of the 4 weeks preceding the medication change.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-02; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Alex deNesnera, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- NAMI NH, Concord, New Hampshire, United States